CLINICAL TRIAL: NCT02266927
Title: An Open-Label, 2-Part, Randomized, Crossover Study to Compare the Bioavailability of Intranasal Administration of 200 and 400 µg of OPTINOSE™ FLUTICASONE With 400 µg of Flonase® (Fluticasone Propionate) Nasal Spray (Part 1), and Intranasal Administration of 200 and 400 µg or 400 µg Alone of OPTINOSE™ FLUTICASONE With 440 µg of Flovent® HFA (Fluticasone Propionate) Inhalation Aerosol (Part 2) (Current Investigation is Part 2 Only)
Brief Title: A Study to Compare the Bioavailability Intranasal Administration of 200 and 400 µg or 400 µg Alone of OPTINOSE™ FLUTICASONE With 440 µg of Flovent® HFA (Fluticasone Propionate) Inhalation Aerosol (Part 2)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Optinose US Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: OPN-FLU-1102
Record Dates: First submitted 2014-10-07; First posted 2014-10-17 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-02

CONDITIONS: Mild to Moderate Asthma
MeSH Terms: interventions — Fluticasone

ARMS (2):
- Flovent® HFA 440µg (Active Comparator): Flovent® HFA (fluticasone propionate) Inhalation Aerosol 440 µg
  Interventions: Drug: Flovent HFA
- OPTINOSE™ FLUTICASONE 400µg intranasal (Experimental): OPTINOSE™ FLUTICASONE, single dose of 400 µg intranasally
  Interventions: Drug: OPTINOSE™ FLUTICASONE

INTERVENTIONS:
Drug: Flovent HFA
  Arms: Flovent® HFA 440µg
Drug: OPTINOSE™ FLUTICASONE
  Arms: OPTINOSE™ FLUTICASONE 400µg intranasal

SUMMARY:
To compare the systemic exposure of a single dose of 400 µg of OPTINOSE FLUTICASONE with 440 µg of Flovent® HFA (fluticasone propionate) Inhalation Aerosol in asthmatic subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects' ages 18 to 55 years, inclusive, at screening.
2. Have a body mass index of 18 to 32 kg/m2, inclusive, and a body weight of not less than 52 kg for males and 45 kg for females.
3. Otherwise healthy mild to moderate asthmatic (Part 2) with no clinically relevant abnormalities in the opinion of the Investigator as determined by medical history, physical examination, blood chemistry, hematology (including complete blood count), serology, urinalysis, vital signs, and ECG performed at screening.
4. History of mild to moderate asthma, diagnosed by a physician, which is well controlled at the present time (no history of sudden or severe asthma exacerbation in the past 12 months).
5. Are unlikely to exacerbate during the study due to seasonal allergen exposure.
6. Able to tolerate withdrawal of their medication for a required period of time.

Exclusion Criteria:

1. Currently have or have a history of disease or dysfunction of the cardiovascular, endocrine, hematologic, neurological, immune, gastrointestinal, genitourinary, musculoskeletal, or other body system that is clinically significant in the opinion of the Investigator.
2. History of smoking or use of nicotine-containing substances within the previous 3 months before screening.
3. Hypersensitivity to fluticasone propionate or any of the excipients found in OPTINOSETM FLUTICASONE or Flovent® HFA (for Part 2).
4. History of extensive nasal and/or sinus surgery.
5. Known nasal obstruction including allergic rhinitis, nasal septal deviations, polyposis, severe mucosal swelling, nasal ulcers, nasal trauma or any other reason.
6. History of acute severe asthma attacks.
7. History of seasonal asthma exacerbation, in which case subjects should be outside the relevant allergen season.
8. Have evidence of any chronic medical conditions other than asthma requiring prescription medications (e.g., hypertension or diabetes).
9. Have used inhaled, intranasal, oral, or injectable corticosteroids within 4 weeks prior to dosing. Subjects should be on stable treatment for at least 1 month prior to withdrawal.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2014-09; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
The ratio of least-squares means of the ln transformed PK parameter AUC0-∞ is the primary endpoint. | Pre-dose and at 0.167, 0.333, 0.5, 0.75, 1, 1.333, 1.667, 2, 2.5, 3, 4, 6, 9, 12, 16, 24, and 36 hours after dosing
  Part 2

CONTACTS AND LOCATIONS:
Overall Officials: Adrian J Stewart, BM, MRCGP, MFPM, Principal Investigator — Celerion
Locations (1):
- Celerion, Belfast, Ireland

REFERENCES:
- [Derived] Messina JC, Offman E, Carothers JL, Mahmoud RA. A Randomized Comparison of the Pharmacokinetics and Bioavailability of Fluticasone Propionate Delivered via Xhance Exhalation Delivery System Versus Flonase Nasal Spray and Flovent HFA Inhalational Aerosol. Clin Ther. 2019 Nov;41(11):2343-2356. doi: 10.1016/j.clinthera.2019.09.013. Epub 2019 Nov 12. PMID 31732149